CLINICAL TRIAL: NCT05265910
Title: A Single-Center, Randomized, Double-Masked, Parallel Study Comparing the Efficacy of Pataday® Once Daily Relief Extra Strength to Claritin® Tablets 24-Hour in Reducing Ocular Itching in Subjects With Allergic Conjunctivitis
Brief Title: A Study Comparing the Efficacy of Pataday® Once Daily Relief Extra Strength to Claritin® Tablets 24-Hour in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andover Research Eye Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-960-0004
Record Dates: First submitted 2021-12-14; First posted 2022-03-04 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pataday® Once Daily Relief Extra Strength and Placebo tablet (Active Comparator): Pataday® Once Daily Relief Extra Strength (olopatadine hydrochloride ophthalmic solution 0.7%) will be administered bilaterally and Placebo tablet will be administered orally (within 5 minutes of eyedrop) at Visits 3 and 4a.
  Interventions: Drug: olopatadine hydrochloride ophthalmic solution 0.7%; Drug: Placebo
- Tears Naturale® II and Claritin® Tablet 24-Hour (Active Comparator): Tears Naturale® II will be administered bilaterally and Claritin® Tablet 24-Hour (loratadine 10 mg) will be administered orally (within 5 minutes of eyedrop) at Visits 3 and 4a.
  Interventions: Drug: loratadine 10 mg; Drug: Tears Naturale

INTERVENTIONS:
Drug: olopatadine hydrochloride ophthalmic solution 0.7% — Pataday® Once Daily Relief Extra Strength (eyedrop)
  Other Names: Pataday® Once Daily Relief Extra Strength
  Arms: Pataday® Once Daily Relief Extra Strength and Placebo tablet
Drug: loratadine 10 mg — Claritin® Tablets 24-Hour (tablet)
  Other Names: Claritin® Tablets 24-Hour
  Arms: Tears Naturale® II and Claritin® Tablet 24-Hour
Drug: Tears Naturale — Tears Naturale® II (eyedrop)
  Other Names: Tears Naturale® II
  Arms: Tears Naturale® II and Claritin® Tablet 24-Hour
Drug: Placebo — Placebo tablet (tablet)
  Other Names: Placebo tablet
  Arms: Pataday® Once Daily Relief Extra Strength and Placebo tablet

SUMMARY:
This is a single-center, randomized, double-masked, parallel study. In this clinical study, the efficacy comparison between Pataday® Once Daily Relief Extra Strength and Claritin® Tablets 24-Hour will be made using the Ora-CAC model, a validated clinical model accepted by regulatory agents for assessing the efficacy of products on the signs and symptoms of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

Each subject must:

1. Be at least 18 years of age at Visit 1 of either gender and any race;
2. Provide written informed consent and sign the HIPAA form;
3. Be willing and able to follow all instructions and attend all study visits;
4. Have a history of ocular allergies and a positive skin test reaction to a seasonal (grass, ragweed, and/or tree pollen) or perennial (cat dander, dog dander, dust mites, cockroach) allergen as confirmed by an allergic skin test conducted at Visit 1 or within the last 24 months;
5. Be able and willing to avoid all disallowed medications for the appropriate washout period and during the study (see exclusion 6);
6. Be able and willing to discontinue wearing contact lenses for at least 72 hours prior to Visit 1 and during the study trial period;
7. (for females capable of becoming pregnant) agree to have urine pregnancy testing performed at screening (must be negative) and exit visit; must not be lactating; and must agree to use a medically acceptable form of birth control throughout the study duration. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
8. Have a calculated best-corrected visual acuity of 0.7 logMAR or better in each eye as measured using an ETDRS chart;
9. Have a positive bilateral post-CAC reaction (defined as having scores of ≥2 ocular itching and ≥2 conjunctival redness) within 10 (±2) minutes of instillation of the last titration of allergen at Visit 1;
10. Have a positive bilateral post-CAC reaction (defined as having scores of ≥2 ocular itching and ≥2 conjunctival redness) for at least two out of the first three time points following the challenge at Visit 2.

Exclusion Criteria:

Each subject must not:

1. Have known contraindications or sensitivities to the use of the investigational product or any of its components; 2. Have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium, history of corneal transplantation or a diagnosis of dry eye); 3. Have had ocular surgical intervention within three (3) months prior to Visit 1 or during the study and/or a history of refractive surgery within the past six (6) months; 4. Have a known history of retinal detachment, diabetic retinopathy, or active retinal disease; 5. Have the presence of an active ocular infection (bacterial, viral, or fungal) or positive history of an ocular herpetic infection at any visit; 6. Use any of the following disallowed medications during the period indicated prior to Visit 1 and during the study: 7 Days

* systemic or ocular H1-antihistamine, H1-antihistamine/mast cell stabilizers, H1-antihistamine-vasoconstrictor drug combinations;
* decongestants;
* monoamine oxidase inhibitors
* all other topical ophthalmic preparations (including artificial tears)
* lid scrubs;
* topical prostaglandins or prostaglandin derivatives
* ocular, topical, or systemic nonsteroidal anti-inflammatory drugs (NSAIDs, including baby aspirin (81 mg)) 14 Days
* inhaled, ocular, topical, or systemic corticosteroids or mast cell stabilizers; 45 Days
* depo-corticosteroids; Note: Currently marketed over-the-counter anti-allergy eye drops (i.e. anti-histamine/vasoconstrictor combination products such as Visine®-A®) may be administered to subjects by trained study personnel at the end of Visits 1, 2 and 4b after all evaluations are completed.

  7. Have any significant illness (e.g. any autoimmune disease requiring therapy, severe cardiovascular disease [including arrhythmias] the investigator feels could be expected to interfere with the subject's health or with the study parameters and/or put the subject at any unnecessary risk (includes but is not limited to: poorly controlled hypertension or poorly controlled diabetes, a history of status asthmaticus, organ transplants, a known history of persistent moderate or severe asthma, or a known history of moderate to severe allergic asthmatic reactions to any of the study allergens; 8. Have received allergy immunotherapy within the last 2 years; 9. Manifest signs or symptoms of clinically active allergic conjunctivitis in either eye at the start of Visits 1, 2, or 3 (defined as the presence of any itching or >1 [greater than 1] redness in any vessel bed); 10. Have a history of glaucoma; 11. Have planned surgery (ocular or systemic) during the trial period or within 30 days after; 12. Have used an investigational drug or medical device within 30 days of the study or be concurrently enrolled in another investigational product trial; 13. Be a female who is currently pregnant, planning a pregnancy, or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Ocular itching 3(±1) minutes post-CAC at Visit 3 | 3(±1) minutes post-CAC on Day 1 (Visit 3)
  Ocular itching evaluated by the subject at 3(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Visit 3.
Ocular itching 3(±1) minutes post-CAC at Visit 4b | 3(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ocular itching evaluated by the subject at 3(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Vi sit 4b.
Ocular itching 5(±1) minutes post-CAC at Visit 3 | 5(±1) minutes post-CAC on Day 1 (Visit 3)
  Ocular itching evaluated by the subject at 5(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Visit 3.
Ocular itching 5(±1) minutes post-CAC at Visit 4b | 5(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ocular itching evaluated by the subject at 5(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Ocular itching 7(±1) minutes post-CAC at Visit 3 | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Ocular itching evaluated by the subject at 7(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Visit 3.
Ocular itching 7(±1) minutes post-CAC at Visit 4b | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ocular itching evaluated by the subject at 7(±1) minutes post-CAC (0-4 on the Ocular Itching scale with 4 being the worst, allowing half unit increments) at Visit 4b.

SECONDARY OUTCOMES:
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Conjunctival Redness | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Conjunctival Redness | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Conjunctival Redness | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Ciliary Redness | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Ciliary Redness | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Ciliary Redness | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Episcleral Redness | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Episcleral redness evaluated by the investigator at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Episcleral Redness | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Episcleral redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Episcleral Redness | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Episcleral redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Chemosis | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Chemosis | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Chemosis | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Eyelid Swelling | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Eyelid Swelling | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Eyelid Swelling | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Tearing | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Tearing | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Tearing | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Rhinorrhea | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Rhinorrhea | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Rhinorrhea | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Nasal Pruritis | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Nasal Pruritis | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Nasal Pruritis | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Ear or Palate Pruritis | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Ear or Palate Pruritis | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Ear or Palate Pruritis | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 3; Nasal Congestion | 7(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal congestion evaluated by the subject (0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 3; Nasal Congestion | 15(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal congestion evaluated by the subject (0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 3; Nasal Congestion | 20(±1) minutes post-CAC on Day 1 (Visit 3)
  Nasal congestion evaluated by the subject 0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 3.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Conjunctival Redness | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Conjunctival Redness | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Conjunctival Redness | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Conjunctival redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Ciliary Redness | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Ciliary Redness | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Ciliary Redness | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ciliary redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Episcleral Redness | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Episcleral redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Episcleral Redness | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Episcleral redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Episcleral Redness | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Episcleral redness evaluated by the investigator (0-4 on the Ocular Redness scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Chemosis | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Chemosis | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Chemosis | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Chemosis evaluated by the investigator (0-4 on the Ocular Chemosis scale with 4 being the worst, allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Eyelid Swelling | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Eyelid Swelling | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Eyelid Swelling | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Eyelid swelling evaluated by the subject (0-3 on the Eyelid Swelling scale with 3 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Tearing | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Tearing | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Tearing | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Tearing evaluated by the subject (0-4 on the Tearing scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Rhinorrhea | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Rhinorrhea | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Rhinorrhea | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Rhinorrhea evaluated by the subject (0-4 on the Rhinorrhea scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Nasal Pruritis | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Nasal Pruritis | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Nasal Pruritis | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal pruritis evaluated by the subject (0-4 on the Nasal Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Ear or Palate Pruritis | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Ear or Palate Pruritis | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Ear or Palate Pruritis | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Ear or palate pruritis evaluated by the subject (0-4 on the Ear or Palate Pruritis scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 7(±1) minutes post-CAC at Visit 4b; Nasal Congestion | 7(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal congestion pruritis evaluated by the subject (0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 15(±1) minutes post-CAC at Visit 4b; Nasal Congestion | 15(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal congestion pruritis evaluated by the subject (0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 4b.
Secondary Efficacy Measures 20(±1) minutes post-CAC at Visit 4b; Nasal Congestion | 20(±1) minutes post-CAC at Visit 4b (24 hours from Visit 4a; Day 15±3)
  Nasal congestion pruritis evaluated by the subject (0-4 on the Nasal Congestion scale with 4 being the worst, not allowing half unit increments) at Visit 4b.

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No